CLINICAL TRIAL: NCT04812054
Title: Improving Quality of Livers Procured for Transplantation From Deceased Donors Using Hypothermic Machine Perfusion
Brief Title: Dual Hypothermic Oxygenated Machine Perfusion in Liver Transplantation Using Allografts From Donors After Brain Death
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1WB1/NCN6; 2019/34/E/NZ5/00433 (Other Grant/Funding Number: National Science Centre, Poland)
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Liver Cirrhosis; Liver Tumor; Liver Transplant Failure and Rejection
Keywords: liver transplantation; machine perfusion; primary non-function
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: Following provision of informed consent, recipients will be randomly assigned in a 1:3 ratio to either hypothermic perfusion group or simple static cold storage group. Randomization will be performed in the blocks of 8 by drawing a sealed envelope by the investigator immediately after organ procurement.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermic oxygenated machine perfusion (Experimental): Allografts will be subject to end-ischemic hypothermic oxygenated perfusion at 12 degrees Celsius through both hepatic artery and portal vein after a period of simple cold storage at 4 degrees Celsius and immediately prior to implantation. The perfusion will last at least 2 hours and the period will be prolonged in case of ongoing hepatectomy, in order to perform graft implantation immediately after perfusion.
  Interventions: Procedure: Hypothermic oxygenated machine perfusion
- Simple cold storage (Active Comparator): Allografts will be stored in perfusate at 4 degrees Celsius from the procurement until implantation.
  Interventions: Procedure: Simple cold storage

INTERVENTIONS:
Procedure: Hypothermic oxygenated machine perfusion — Hypothermic oxygenated perfusion using a Liver Assist device (Organ Assist, Groningen, the Netherlands). Temperature of the perfusate will be set to 12 degrees Celsius. Dedicated cannulas will be placed in the aorta for arterial perfusion and in the portal vein for portal perfusion. Pressure will be set at 25 mmHg for arterial line (pulsatile flow, 30 mmHg systolic pressure and 20 mmHg diastolic pressure, 60 beats per minute) and 3 mmHg for portal line (continuous flow). 100% oxygen will be supplied to the oxygenators with a flow of 500 ml / min or higher, in order to achieve pO2 of at least 450 mmHg.
  Other Names: DHOPE
  Arms: Hypothermic oxygenated machine perfusion
Procedure: Simple cold storage — Following back-table preparation, the allograft will either be transferred to the operating room for implantation or stored in preservation solution at 4 degrees Celsius in a refrigerator
  Arms: Simple cold storage

SUMMARY:
This will be a randomized study on the effects of hypothermic oxygenated machine perfusion in patients undergoing liver transplantations from donors after brain death with allocation of patients to either end-ischemic hypothermic oxygenated machine perfusion group (at least 2 hours of allograft perfusion at 12 degrees Celsius though hepatic artery and portal vein prior to implantation) or simple cold storage group in a 1:3 ratio. The primary outcome measure of the study will be model for early graft dysfunction (MEAF) score. A total number of 104 patients, including 26 in the hypothermic perfusion group and 78 in simple cold storage group will be included. Data on potential risk factors for worse allograft function and increased ischemia-reperfusion injury will be collected perioperatively. Circulating levels of proinflammatory cytokines (IL-2, IL-10, TNFα), nuclear damage (HMGB-1, 8-OHdG), serum activity of transaminases, gamma-glutamyl-transpeptidase, bilirubin concentration, and INR will be assessed in the perioperative period. Wedge allograft biopsies will be performed 90 minutes post-reperfusion to evaluate activation of innate immunity (TLR4), activation of endothelium (vWF, P-selectin), hepatocyte necrosis, hepatocyte apoptosis (TUNEL assay), ATP content, and oxidative damage (malondialdehyde content). Further, wedge biopsies will be performed at the end of simple cold storage and at the beginning and after two hours of perfusion to determine steatosis and ATP content. During the perfusion, perfusate samples will be periodically tested for lactate, sodium, and potassium concentration, CO2 partiall pressure, and flavin mononucleotide concentration. Patients will be closely monitored in the postoperative period for allograft function and secondary end-points: 2-year recipient and graft survival, 2-year incidence of biliary complications, and 90-day complication rate. Both groups will be compared with respect to the primary and secondary end-points, circulating levels of IL-2, IL-10, TNFα, HMGB-1, 8-OHdG, activity of transaminases and gamma-glutamyl-transpeptidase, and findings in post-reperfusion allograft biopsies. Further, changes of hepatic steatosis and hepatic ATP content during perfusion will be evaluated, and the results of perfusate analyses will be tested as predictors of allograft function in the post-transplant period.

DETAILED DESCRIPTION:
This will be a parallel, randomized controlled study on the effects of end-ischemic hypothermic oxygenated machine perfusion in liver transplantations from donors after brain death. Patients will be randomized to either hypothermic perfusion or simple cold storage (1:3 ratio). The primary end-point will be model for early graft dysfunction (MEAF) score, a recently validated continuous measure of allograft function in the early period after liver transplantation, calculated using serum alanine transaminase (ALT) activity, international normalized ratio for prothrombin time (INR), and serum bilirubin concentration within 3 first postoperative days. In the original study, the mean MEAF score was 5.01 with a standard deviation of 1.99. The primary hypothesis of this study is reduction of the mean MEAF score from 5 to 3.5 using hypothermic oxygenated machine perfusion. With the thresholds for type I error of 0.05 and power of 0.90, respectively, 1:3 allocation ratio, and a standard deviation of 1.99, the number of patients required to detect such difference is 26 in the hypothermic perfusion group and 78 in the simple cold storage group (104 in total). The inclusion criteria will comprise age >18 years, deceased-donor liver transplantation, and provision of informed consent. Exclusion criteria will comprise donation after cardiac death and either reduced or split graft. Secondary outcome measures will include 2-year recipient and graft survival, 2-year incidence of biliary complications, and complications in the 90-day postoperative period classified by type and their severity according to the Clavien-Dindo grading system.

Following provision of informed consent, recipients will be randomly assigned in a 1:3 ratio to either hypothermic perfusion group or simple static cold storage group. In the hypothermic perfusion group, allografts will be subject to end-ischemic hypothermic oxygenated perfusion at 12 degrees Celsius through both hepatic artery and portal vein after a period of simple cold storage at 4 degrees Celsius and immediately prior to implantation. The perfusion will last at least 2 hours and the period will be prolonged in case of ongoing hepatectomy, in order to perform graft implantation immediately after perfusion. Two wedge allograft biopsies will be performed at the beginning and after 2 hours of perfusion for the assessment of micro- and macrovesicular steatosis and ATP content. Samples of the perfusate will be taken at the beginning and every 30 minutes for the assessment of sodium, potassium, and lactate concentration, CO2 partial pressure, and FMN. Perfusate temperature, portal and arterial flow, and portal and arterial resistance will be closely monitored during the procedure. In the simple cold storage group, the allografts will be stored in perfusate at 4 degrees Celsius from the procurement until implantation. At the end of simple cold storage, a wedge biopsy will be taken for the assessment of micro- and macrovesicular steatosis and ATP content. In both groups during the back-table procedure, the allograft will be flushed with 1 litre of perfusate through the portal vein. At the end of flushing, a sample of perfusate will be taken from the right hepatic vein for assessment of FMN and lactate concentration.

In both groups, clinical, anthropometric, and laboratory pre-transplant data will be collected. This includes: indication for transplantation, Child-Turcotte-Pugh classification, presence of hepatitis B and C virus infection, model for end-stage liver disease (MELD) score (without exception points), patient weight, height, body mass index, and waist circumference, serum bilirubin, creatinine, glucose and albumin concentration, INR, and serum activity of transaminases. Relevant donor and procurement data will be collected, including donor age, height, body mass index, cause of death, ethnicity, serum sodium and bilirubin concentration, serum activity of transaminases, INR, and extraction time. Donor risk index will be calculated in every case. Duration of cold ischemia and several intraoperative parameters will be collected, including: duration of warm ischemia, intraoperative transfusions, serum sodium and potassium changes, occurrence of post-reperfusion syndrome, and duration of operation. A wedge biopsy will be performed in all patients 90 minutes after portal reperfusion for histological assessment of ischemia-reperfusion injury (Suzuki score), apoptosis, endothelial activation (vWF and P-selectin), activation of innate immunity (TLR4) , oxidative injury (MDA), and ATP content. Blood samples will be collected immediately prior to reperfusion, 90 minutes after reperfusion, and at first postoperative day for the assessment of proinflammatory cytokines (TNFα, IL-2, IL-10), nuclear damage (HMGB1, 8-OHdG) and hepatocyte and cholangiocyte injury (transaminases and GGT activity). Following transplantation, all patients will be strictly followed according to the centre protocol with the assessment of serum activity of transaminases and GGTP, bilirubin and creatinine concentration, and INR twice daily within the first 3 postoperative days and daily or once every 2-3 days (according to the clinical assessment) thereafter. All complications occurring during the 90-postoperative period will be recorded, including primary non-function, early allograft dysfunction, biliary leaks, rejection episodes, and vascular complications. After hospital discharge, patients will be followed-up according to the center protocol with regular appointments in the outpatient clinic, every 2 weeks within first 2 months post-transplantation, every month up to 6 months, every 2-3 months up to 1 year, and every 3-6 months thereafter. Occurrence of all complications, particularly biliary complications, will be recorded. Both groups will be compared with respect to primary and secondary outcome measures, other pre-defined clinical outcomes, allograft injury and ATP content before implantation, and signs of ischemia-reperfusion injury, oxidative damage, apoptosis, ATP content, activation of innate immunity, and endothelial activation in allograft biopsies after reperfusion. Comparisons will also include pro-inflammatory cytokine release, circulating markers of nuclear injury, and other laboratory markers of allograft function and injury. Analyses of perfusate samples and allograft biopsies obtained before and after reperfusion is planned in order to determine both the impact of hypothermic perfusion on hepatic ATP content and mitochondrial injury (FMN). Further, results of perfusate analyses (particularly FMN) will be evaluated for potential association with clinical outcome measures, results of post-reperfusion allograft biopsies assessment, and serum markers of allograft function, injury, and inflammatory response in order to determine its role in pre-transplant assessment of allograft viability.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* deceased-donor liver transplantation
* provision of informed consent

Exclusion Criteria:

* donation after cardiac death
* either reduced or split graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Model for early graft dysfunction score | 3 days
  Continuous measure of allograft function in the early period after liver transplantation, calculated using serum alanine transaminase (ALT) activity, international normalized ratio for prothrombin time (INR), and serum bilirubin concentration within 3 first postoperative days

SECONDARY OUTCOMES:
Recipient survival | 2 years
  Recipient survival over 2-year follow-up
Graft survival | 2 years
  Graft survival (retransplantation or death) over 2-year follow-up
Biliary complications | 2-years
  Incidence of biliary complications (bile leaks, strictures) over 2-year follow-up
Postoperative complications | 90 days
  Complications in the 90-day postoperative period classified by type and their severity according to the Clavien-Dindo grading system

OTHER OUTCOMES:
Cytokine release in the perioperative period | 1 day
  Serum levels of IL-2, IL-10, TNFα, HMGB-1, and 8-OHdG before reperfusion, 90 minutes after reperfusion, and 24 hours after reperfusion
Allograft ischemia-reperfusion injury | 90 minutes
  Suzuki score in wedge allograft biopsy 90 minutes after reperfusion
Hepatocyte apoptosis in the allograft | 90 minutes
  TUNEL assay in wedge allograft biopsy 90 minutes after reperfusion
Endothelial activation in the allograft | 90 minutes
  vWF and P-selectin staining in wedge allograft biopsy 90 minutes after reperfusion
Activation of innate immunity in the allograft | 90 minutes
  TLR4 staining in wedge allograft biopsy 90 minutes after reperfusion
Oxidative injury of the allograft | 90 minutes
  MDA assay in wedge allograft biopsy 90 minutes after reperfusion
Allograft ATP content | 90 minutes
  ATP content in wedge allograft biopsy 90 minutes after reperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Michal Grat, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of General, Transplant and Liver Surgery, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Information will be available from the investigators upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from the investigators upon reasonable request following the publication of final article reporting on all primary and secondary outcome measures
Access Criteria: Requests should be addressed to the principal investigator

REFERENCES:
- [Derived] Grat M, Morawski M, Zhylko A, Rykowski P, Krasnodebski M, Wyporski A, Borkowski J, Lewandowski Z, Kobryn K, Stankiewicz R, Stypulkowski J, Holowko W, Patkowski W, Mielczarek-Puta M, Struga M, Szczepankiewicz B, Gornicka B, Krawczyk M. Routine End-ischemic Hypothermic Oxygenated Machine Perfusion in Liver Transplantation From Donors After Brain Death: A Randomized Controlled Trial. Ann Surg. 2023 Nov 1;278(5):662-668. doi: 10.1097/SLA.0000000000006055. Epub 2023 Jul 27. PMID 37497636